CLINICAL TRIAL: NCT06381687
Title: A Movement and Music Programme in Early Childhood Education and Care to Promote Physical Activity, Gross and Fine Motor and Musical Skills: The MoviMusi Study Protocol
Brief Title: A Movement and Music Programme in Early Childhood Education and Care (The MoviMusi Study Protocol)
Acronym: MOVIMUSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Vladimir Martínez Bello, Senior Lecturer, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-3118978; PID2022-141095NB-I00 (Other Grant/Funding Number: Spanish Ministry of Science, Innovation and Universities)
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Fundamental Motor Skills; Physical Activity; Music Intervention
Keywords: Early Childhood; Movement behaviors; Gross and fine motor skills
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The allocation of ECECs to the intervention versus control group will be randomised in a blinded procedure at the end of the first year, following the baseline assessment. Once ECEC centres meeting the selection criteria are identified, they will be randomised to one of the trial arms.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention: characteristics of the movement and music programme (Experimental): A multi-component, multi-level programme (MoviMusi) will be designed and implemented in each city by the 12 ECEC centres in the intervention group. The intervention programme will start after baseline measurements and it will be implemented during 12 months. Accompanied by members of the intervention team, the educational community will be empowered to identify areas for improvement and make the necessary changes in their centres. In addition, the intervention programme will aim to address the main barriers and facilitators identified during the first year (baseline assessment) in relation to movement and music curricular practices.
  Interventions: Behavioral: A multi-component, multi-level programme (MoviMusi)
- Control group (No Intervention): In the three cities, 12 ECEC institutions will participate in the control group. The centres will follow their usual curricular programme and will be visited to identify the curricular movement and music practices they are implementing, to assess the quality of the school environment and to measure PA, gross and fine motor skills, and music skills at baseline and at the end of the study.

INTERVENTIONS:
Behavioral: A multi-component, multi-level programme (MoviMusi) — The MoviMusi program will be designed and implemented in each city by the 12 ECEC centres in the intervention group. In addition, the intervention programme will aim to address the main barriers and facilitators identified during the first year (baseline assessment) in relation to movement and music curricular practices. The programme will have three axes:
  (1) Training. Educators and families will actively participate in a series of seminars and training workshops on the promotion of PA as a healthy behaviour and the use of music as a didactic resource to strengthen holistic education both inside and outside ECEC. (2) Participation. Each ECEC institution will be supported as they design a movement and music programme to offer children better opportunities to learn about the body, its possibilities of action, and musical skills.(3) Implementation. The specific actions of the MoviMusi Programme will be put into practice in each ECEC institution.
  Arms: Experimental intervention: characteristics of the movement and music programme

SUMMARY:
The early childhood education and care (ECEC) environment is an important setting for providing children with daily opportunities for movement and music, supporting holistic child development in the early years. To date, there are no studies evaluating the implementation of a holistic programme in the ECEC context in the areas of movement behaviour, motor, and musical skills. The main aim is to examine the impact over time of a holistic movement and music programme on correlates of movement behaviour, gross and fine motor skills, and musical skills in young children (1-3 years). The secondary aims are to examine the impact of the movement and music programme on the perceptions of the educational community, as well as the barriers and facilitators they perceive in the process of baseline assessment, construction, and implementation of the movement and music programme in their own ECEC community. This cluster-randomised controlled trial (intervention and control groups) with public ECEC centres will be performed over a 24-month period. Baseline measurements will be taken in the first year of the project, and the longitudinal evaluation of the implementation of the movement and music programme in the second year. educational community's perceptions about the barriers and facilitators associated with the correlates of movement behaviour will be taken into account, as will the results of the assessment of gross and fine motor and musical skills identified in the first year of the project, with a special focus on the structured and unstructured opportunities for movement and music both in the ECEC settings and at home. This research project aims to fill a knowledge gap during a period of childhood that has rarely been explored, either nationally or internationally (1-3 years), and to position movement and music teaching practices as key contexts in the curriculum development of infant and toddler education.

DETAILED DESCRIPTION:
ECEC settings are important determinants of children´s behaviour. Ecological models help to contextualise and explain how the different environments in which children interact on a daily basis (school, home, and peer relations) have the capacity to influence childrens development. To date, there are no studies evaluating the implementation of a holistic programme in the ECEC context in the areas of movement behaviour, motor, and musical skills. A pending line of research is the identification of the key correlates of changes in movement behaviour throughout the early years, which would generate knowledge crucial to developing policy interventions that promote general wellbeing in young children. Thus, this study focuses on the importance of home and ECEC settings in the development of movement behaviour through a critical analysis of how curricular practices can be more effective in influencing childrens holistic development.

Aims The main aim is to examine the impact over time of a holistic movement and music programme on correlates of movement behaviour, gross and fine motor skills, and musical skills in young children (1-3 years). The secondary aims are to examine the impact of the movement and music programme on the perceptions of the educational community, as well as the barriers and facilitators they perceive in the process of baseline assessment, construction, and implementation of the movement and music programme in their own ECEC community.

Hypotheses The research set out to test the following hypotheses: 1. Girls and boys (1-2 years) will perform the same amount of PA during the school day. 2. The implementation of a music and movement intervention programme will increase children´s PA during the school day. 3. The music and movement intervention programme will have an impact on higher levels of childrens GMS as well as a variety of musical processes in the intervention group. 4. The ECEC community will be actively involved in the co-creation process of the movement and music intervention programme.

ELIGIBILITY:
Inclusion Criteria:

* Young children aged 14 to 22 months.
* Regularly attending the Early Childhood Education and Care centre.
* Parents giving informed consent.

Exclusion Criteria:

* Young children not attending more than two days to centre.
* Young children attending only half part of the day.

Ages: 14 Months to 22 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 312 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity | At baseline and 12 months
  Accelerometry (Actigraph model) will be used to objectively assess physical activity. Children will wear an accelerometer for one week (weekend included) during ECEC hours. Accelerometer data will be downloaded and converted to 15-s epoch files using ActiLife software (version 6.4, ActiGraph Inc, Pensacola, FL, USA).
Sleep time | At baseline and 12 months
  Sleep time wil be measured by parental report.
Motor skills | At baseline and 12 months
  Participants' motor skills will be assessed using the Peabody Developmental Motor Scales, 3rd edition. The PDMS-3 is a standardized instrument to assess both gross and fine motor skills.
Musical skills | At baseline and 12 months
  Musical skills will be assessed using a observational approach based on the five fundamental musical processes (listening, singing, instrumental interpretation, improvisation/composition and movement).
Sedentary time | At baseline and 12 months
  Accelerometry (Actigraph model) will be used to objectively assess sedentary time. Children will wear an accelerometer for one week (weekend included) during ECEC hours. Accelerometer data will be downloaded and converted to 15-s epoch files using ActiLife software (version 6.4, ActiGraph Inc, Pensacola, FL, USA).

SECONDARY OUTCOMES:
For young children, the first secondary outcome measure is physical activity and sedentary time during unstructured and structured physical activity opportunities. | At baseline and 12 months
  Accelerometry (Actigraph model) will be used to objectively assess sedentary time. Children will wear an accelerometer during unstructured and structured physical activity opportunities.
For young children, the second secondary outcome measure will be the play patterns during unstructured outdoor free play. | At baseline and 12 months
  The OSRAC-P is a direct observation system designed to collect information about children's physical activity and the contextual circumstances surrounding it (Brown et al., 2006).
For ECEC educators, the first secondary outcome will be the perceived barriers and facilitators for the inclusion of movement and music as curricular practices in the ECEC institution. | At baseline and 12 months
  In each ECEC setting, educators will participate in focus groups to gather their perceptions about the place and purpose of movement and music practices in their classrooms.
For ECEC educators, the second secondary outcome will be the perceived impact of the implementation of the movement and music program. | At baseline and 12 months
  In each ECEC setting, educators will participate in focus groups, to gather their perceptions about the place and purpose of movement and music practices in their classrooms.
For families, the first secondary outcome is the perceived barriers and facilitators to PA in young children. | At baseline and 12 months
  Barriers to active commuting will be assessed using an adapted version of the BATACE scale (BArreras en el Transporte Activo al Centro Educativo in Spanish, translated as: barriers to active transport to educational centres) for preschool and toddler parents.
For families, the second secondary outcome is the perceived barriers and facilitators to the inclusion of music at home. | At baseline and 12 months
  In each ECEC setting, families will participate in focus groups, in order to identify their perceptions of barriers and facilitators to movement and music practice outside of school hours.
For families, the third secondary outcome are the means of transport to ECEC settings and barriers to active comm | At baseline and 12 months
  The modes of transport used for commuting to and from the ECEC centre will be evaluated through a questionnaire.
For families, the fourth secondary outcome is the habitual perceived PA and sedentary behaviour in the child's home environment. | At baseline and 12 months
  The Preschool-aged Children's PA Questionnaire (Pre-PAQ) is a questionnaire designed to measure habitual PA and sedentary behaviour in the child's home environment.
For families, the fifth secondary outcome is the perceived barriers and facilitators to PA in young children. | At baseline and 12 months
  Barriers to active commuting will be identified also by a qualitative analysis in focus groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
The Spanish government has given us a grant without taking into account this policy.

REFERENCES:
- [Background] undefined
- [Background] Gubbels JS, Van Kann DHH, Cardon G, Kremers SPJ. Activating Childcare Environments for All Children: the Importance of Children's Individual Needs. Int J Environ Res Public Health. 2018 Jul 3;15(7):1400. doi: 10.3390/ijerph15071400. PMID 29970831
- [Background] Carson V, Draper CE, Okely A, Reilly JJ, Tremblay MS. Future Directions for Movement Behavior Research in the Early Years. J Phys Act Health. 2023 Dec 18;21(3):218-221. doi: 10.1123/jpah.2023-0679. Print 2024 Mar 1. No abstract available. PMID 38109880